CLINICAL TRIAL: NCT03389997
Title: Assessement of Viral Shedding Duration After a Respiratory Tract Infection in Oncology and Hematology Patients
Acronym: ONCOVIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ONCOVIR
Record Dates: First submitted 2017-12-21; First posted 2018-01-04 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Respiratory Tract Viral Infection
Keywords: respiratory tract infections; virus shedding; cancer; Immunocompromised Host
MeSH Terms: conditions — Respiratory Tract Infections; Neoplasms

STUDY DESIGN:
Intervention Model Description: Iterative nasal swabs will be performed to screen for virus shedding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: nasal swabs — Iterative nasal swabs will be performed to screen for virus shedding

SUMMARY:
The purpose of this study is to assess the duration of the viral shedding in hematology and oncology patients after a respiratory tract viral infection. This duration has not been much studied in that population whereas it is probably longer than that in immunocompetent patients. Thereby it may be a source of transmission amongst these immunocompromised patients.

DETAILED DESCRIPTION:
The development of multiplex polymerase chain reaction (PCR) tests has greatly improved the diagnosis of respiratory tract viral infections by increasing its sensitivity and the diversity of viral species detected. However, there are few data concerning respiratory tract viral infections amongst hematology and oncology patients. Especially, the duration of viral shedding following an infection has not been much studied whereas it is a source of inter-individual transmission between immunocompromised patients who are more likely to develop severe disease.

Studies conducted so far concerned mainly hematology patients. They have shown that viral carriage could last up to one month and a half in some patients with hematological malignancy.

The aim of this study is to determine the duration of the viral shedding in patients from hematology and oncology units after a respiratory tract viral infection for the ten main viruses involved in order to better manage these infections and to better prevent their transmission.

ELIGIBILITY:
Inclusion Criteria:

* Patient with solid organ cancer or haematological malignancy with or without chemotherapy
* Having symptoms of upper and/or lower respiratory tract infection
* Virus detected by PCR in nasal sample
* Signature of consent

Exclusion Criteria:

* Hematological stem cell and solid organ recipients
* No health insurance
* protected people

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Nasal carriage of virus after a viral respiratory tract infection | Up to 1 year
  Iterative nasal swab to assess the duration of that carryiage

SECONDARY OUTCOMES:
Prevalence of upper and lower respiratory tract infections | 2 years
Prevalence of viral coinfections | 2 years
Prevalence of bacterial coinfections | 2 years
transmission of respiratory tract viral infections by relatives | 2 years
  with a survey filled by the patient
respiratory complications due to respiratory tract viral infections | 2 years
extra-pulmonary symptoms due to respiratory tract viral infections | 2 years
effect of influenza vaccine on viral shedding | 2 years
risk factors to do severe form of respiratory tract infection | 2 years
nosocomial transmission of respiratory tract viral infection | 2 years
delay of chemotherapy due to respiratory infection | 2 years
survival after a respiratory tract viral infection | 30 days
TTV viral load as a marker of immunodepression in oncology and hematology patients | 2 years
  TTV viral load at each visit
Correlation between TTV viral load and duration of viral shedding and severity of respiratory tract infection | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: France CAZENAVE-ROBLOT, MD,PhD, Principal Investigator — CHU of POITIERS
Locations (1):
- University Hospital of Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: No